CLINICAL TRIAL: NCT04035629
Title: A Prospective Study of Hyperpolarized 129 Xe MRI in in a Pediatric Population With Bronchopulmonary Dysplasia
Brief Title: 129Xe MRI in Pediatric Population With BPD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not secure funding.
Sponsor: Xemed LLC (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-014532
Record Dates: First submitted 2019-05-31; First posted 2019-07-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: BPD
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hyperpolarized 129Xe MRI for lung diagnosis (Experimental): All subjects will undergo hyperpolarized 129-Xenon MR imaging (HP MRI) and conventional proton MR imaging of lung.
  Interventions: Combination Product: MagniXene, hyperpolarized 129Xe MRI

INTERVENTIONS:
Combination Product: MagniXene, hyperpolarized 129Xe MRI — All subjects will undergo hyperpolarized 129-Xenon MR imaging (HP MRI) and conventional proton MR imaging of lung. Hyperpolarized 129Xe gas is prepared in a process termed spin-exchange optical pumping.
  Xenon is highly lipophilic and therefore soluble in blood and tissue, making it an excellent tool for imaging the gas in both the air spaces (gas-phase imaging) and dissolved in the lung parenchyma (dissolved-phase imaging). This solubility in combination with xenon's chemical shift properties, results in the possibility of quantifying pulmonary gas exchange and gas transport within the parenchyma.
  Additionally, previous images and lung function tests will be reviewed to compare findings and evaluate if there is a correlation between the obtained results.

SUMMARY:
Hyperpolarized (HP) gas magnetic resonance imaging (MRI) of the lungs offers additional information that cannot be obtained with CT scan, the current gold standard for imaging this disorder. As a nonionizing technique, MRI is an ideal modality for pulmonary imaging; in particular in the infant and pediatric population. Nevertheless, due to the low proton density of the lung parenchyma (only ~20% that of solid tissues), numerous air-tissue interfaces that lead to rapid signal decay, and cardiac and respiratory sources of motion that further degrade image quality , MRI has played a limited role in the evaluation of lung pathologies. In this setting, HP gas (using 129Xe) MRI may play a role in helping determine the regional distribution of alveolar sizes, partial pressure of oxygen, alveolar wall thickness, and gas transport efficiency of the microvasculature within the lungs of infants with a diagnosis of bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
The most common respiratory complication of preterm birth, bronchopulmonary dysplasia (BPD), defined by a clinically assessed need for supplemental oxygen support at 36 weeks post-menstrual age, has actually increased in incidence as advancements in clinical respiratory care have improved initial survivability for very premature neonates. However, the burden of pulmonary disease continues beyond the NICU; the survivors are at greater risk for respiratory-related rehospitalization and diminished pulmonary capacity. Pulmonary imaging of the neonate has been limited to the clinical assessment of acute changes in respiratory status. The most widely accessible clinical imaging modalities, radiograph and computed tomography (CT), have significant limitations. Chest radiograph's sensitivity in the acute setting is limited because patients with significant respiratory dysfunction may exhibit only minor radiographic abnormalities, and although CT is considered the gold standard for clinical pulmonary imaging, it is not widely implemented because neonates may require sedation, especially for high-resolution CT, and are especially vulnerable to damage from ionizing radiation. Furthermore, CT is not appropriate for longitudinal assessment because of the link between serial radiation exposure and increased cancer risk.

As a nonionizing technique, magnetic resonance imaging (MRI) is an ideal modality for pulmonary imaging; in particular in the infant and pediatric population. Nevertheless, due to the low proton density of the lung parenchyma (only ~20% that of solid tissues), numerous air-tissue interfaces that lead to rapid signal decay, and cardiac and respiratory sources of motion that further degrade image quality, MRI has played a limited role in the evaluation of lung pathologies. Pulmonary MRI of the neonate is additionally confounded by small patient size and the delicate nature of transporting a NICU patient to the scanner. To overcome these limitations, the use of inhaled, hyperpolarized (HP) noble gases such as helium-3 (3He) and xenon-129 (129Xe) has come into play. Filling the air spaces within the lungs with either of these HP gases provides enough signal and contrast to obtain quality images on MRI.

There has been extensive work with HP 3He MRI in both the adult and pediatric population, but this gas is in extremely limited supply, making it increasingly expensive. 129Xe, on the other hand, is part of the atmosphere and as such does not suffer from supply constraints. Also, xenon dissolves in the lung tissue and blood, a process that is associated with characteristic shifts in the resonance frequency of 129Xe. As a result, the uptake and subsequent transport of 129Xe gas by the pulmonary circulation can be monitored, quantified and analyzed with regard to lung function at a temporal and spatial resolution that is infeasible with any other existing non-invasive modality.

In this study, the lung function in up to 30 infant subjects will be evaluated using HP 129Xe MRI. The subjects will be intubated and sedated neonates with known diagnosis of BPD. Although these subjects have lung disease and may be chronically intubated, they are stable clinically and not acutely ill decreasing the overall risk. When inhaled, 129Xe can be imaged within the lung parenchyma. Using a set of specialized MRI pulse sequences, the diffusion and gas-exchange properties of 129Xe in the lungs of these subjects will be evaluated. This will enable the investigators to determine the regional distribution of alveolar sizes, partial pressure of oxygen, alveolar wall thickness, and gas transport efficiency of the microvasculature within the lung. Each participant will be imaged once using HP 129Xe MRI along with the additional routine proton MRI sequences to further evaluate the structure, volume, and perfusion of the lung parenchyma.

The overall goal of this study is to develop improved quantitative imaging-based lung function parameters to evaluate BPD and determine the phenotypical variants of BPD using HP MRI. HP gas MRI offers additional information that cannot be obtained with CT, the current gold standard for imaging this disorder. Further, MRI offers the advantage of non-ionizing radiation, which is all the more important in the pediatric population particularly within this population who may getting repeat CT examinations throughout their lifetime. Although older children and adults may also benefit from this technology, the improved imaging and phenotyping of BPD will hopefully guide further treatment refinements of this complex disorder.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU at the Children's Hospital of Philadelphia with bronchopulmonary dysplasia who are followed by the Chronic Lung Disease Program.
* Subjects mechanically ventilated either via and endotracheal tube or via a tracheostomy.
* Subjects already receiving sedation as part of clinical care.

Exclusion Criteria:

- Infants whom the primary care team deems to be unstable for transport to MRI

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze 129Xe MRI ventilation maps for regions of abnormal ventilation. | 2 years
  129Xe MRI can reveal unventilated regions of the lungs where the gas cannot reach after being inhaled due to restrictions of the airways.
Analyze 129Xe MRI ADC maps and check for regions of deviations from literature reported normal values. | 2 years
  Apparent diffusion coefficient (ADC) maps are extracted 129Xe MRI from a single breath-hold pulse sequence. Reference values for healthy lungs are available in literature.
Analyze oxygen partial pressure (PAO2) maps extracted from 129Xe MRI | 2 years
  Oxygen partial pressure (PAO2) maps can be extracted from 129Xe MRI maps in a single breath-hold. Regions of the lungs that show abnormal PAO2 values are susceptible of improper ventilation or gas exchange.
Analyze gas exchange and transport coefficient maps and global values as extracted from 129Xe MRI. | 2 years
  Xenon is soluble in lung tissue and blood and can be used for characterizing gas exchange properties at the alveolar level.

SECONDARY OUTCOMES:
Compare 129Xe biometrics to structural magnetic resonance imaging of the lung and clinically available CT and CT angiograms. | 2 years
  Parameters extracted from 129Xe MRI will be studied for correlations with standard proton MRI of the lung and clinically available CT and CT angiograms.
Correlate 129Xe MRI derived ventilation/perfusion (V/Q) measures to a standard clinically used measure of V/Q. | 2 years
  Gas exchange maps as extracted from 129 Xe MRI will be studied for correlations with standard of care clinically measures of V/Q, typically available as medical records.
Correlate 129Xe biometrics to right and left pulmonary arterial flow. | 2 years
  Parameters extracted from 129 Xe MRI as global measures as well as 2D/3D maps will be checked for right lung to left lung variations.

CONTACTS AND LOCATIONS:
Overall Officials: David M Biko, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No